CLINICAL TRIAL: NCT06807632
Title: Phase I Study of Valemetostat and Atezolizumab as Maintenance Therapy for Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Valemetostat in Combination With Atezolizumab in People With Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-290
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: Valemetostat; Atezolizumab; Maintenance therapy; 24-290
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: This is a single institution phase 1 study to assess the safety of valemetostat when used in combination with atezolizumab for the treatment of extensive-stage SCLC patients.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valemetostat in Combination With Atezolizumab (Experimental): This is a single institution phase 1 study to assess the safety of valemetostat when used in combination with atezolizumab for the treatment of extensive-stage SCLC patients. We will begin enrollment at a valemetostat dose of 150 mg once daily (dose level 1), with atezolizumab given per standard of care 1680 mg intravenously every four weeks. The study will have two phases, a dose finding phase and an expansion phase.
  Interventions: Drug: Valemetostat; Drug: Atezolizumab

INTERVENTIONS:
Drug: Valemetostat — Dose level -1 100 mg po once daily
  Dose level 1 150 mg po once daily
  Dose level 2 200 mg po once daily
Drug: Atezolizumab — 1680 mg IV q4weeks

SUMMARY:
This study will test whether valemetostat in combination with atezolizumab is a safe treatment that causes few or mild side effects in people with extensive-stage small cell lung cancer (SCLC). The researchers will test different doses of valemetostat to find the highest dose that causes few or mild side effects in participants. After the dose is found, researchers will test it in a new group of participants to learn more about the safety of the study treatment and see if it is an effective treatment for extensive-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Ability to comply with the study protocol as per the investigator's judgment
* Age ≥ 18 years at the time of signing the ICF
* Life expectancy ≥ 12 weeks
* ECOG performance status 0 or 1
* Pathologically confirmed diagnosis of newly diagnosed extensive-stage small cell lung cancer. Patients with a diagnosis of combined small cell lung cancer with other histologies may be considered for inclusion if the predominant histology is SCLC and only after discussion with the study PI.
* Radiographically documented RECIST version 1.1 stable disease, partial or complete response after initial treatment with a platinum doublet regimen in combination with atezolizumab for 4 cycles. It is acceptable to have no measurable disease at the start of this study.
* Must be able to begin therapy within 4 weeks of completing the fourth cycle of chemotherapy and immunotherapy.
* Adequate hematologic and end-organ function, as defined by the following laboratory test results obtained within 14 days prior to initiation of study treatment. Transfusion (red blood cell or platelet) or granulocyte-colony stimulating factor (G-CSF) administration is not allowed within 2 weeks prior to screening laboratory tests:

  o Adequate bone marrow function as defined by:
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1500/µL)
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100 x 10^9/L o Adequate renal function as defined by:
* Creatinine clearance ≥ 30 mL/min as calculated using the Cockcroft-Gault equation

  o Adequate hepatic function as defined by:
* AST, ALT, and alkaline phosphatase (ALP) ≤ 3 x ULN with the following exception:
* Patients with documented liver metastases: AST, ALT and ALP ≤ 5 x ULN

Exclusion Criteria:

* Any active uncontrolled systemic diseases or other medical conditions considered to be poorly controlled by the investigator including but not limited to bleeding diatheses, that could in the investigator's opinion, potentially interfere with completion of study procedures or interpretation of study outcomes.
* Patients who receive consolidative chest radiation after completion of initial chemotherapy and immunotherapy.
* Symptomatic CNS metastases
* Patients with treated CNS metastases are allowed on the study if their clinical symptoms are adequately controlled and the daily dose of steroid use is equivalent to or less than 10 mg of prednisone.
* Receiving concomitant treatment with a moderate or strong inducer of CYP3A within 14 days of first receipt of valemetostat o Consumption of herbs/fruits that may have an influence on PK of valemetostat (strong CYP3A inhibitors or inducers) such as St. John's wort, star fruit, Seville orange or Seville orange-containing foods and beverages, grapefruit or grapefruit-containing food or beverages should be avoided from 14 days prior to the start of the study and throughout the entire study.

Prior exposure to valemetostat or other inhibitors of enhancer of zeste homologue-2 (EZH2)

* Refractory nausea and vomiting, malabsorption, biliary shunt, significant bowel resection, or any other condition that significantly affects gut motility or absorption and would preclude adequate absorption of valemetostat in the opinion of the treating physician and/or PI.
* Currently receiving radiation therapy, or who have received radiation within 2 weeks prior to the initiation of study treatment, or who plan to receive radiation therapy within the safety evaluation period for dose-limiting toxicity during Cycle 1.
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE version 5.0, Grade ≤ 1 or baseline.

  o NOTE: Participants may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to Grade >2 for at least 3 months prior to enrollment and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, comprised of the following:
* Chemotherapy-induced neuropathy
* Residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include:
* Hypothyroidism/ hyperthyroidism
* Type I diabetes
* Hyperglycemia
* Adrenal insufficiency
* Adrenalitis
* Skin hypopigmentation (vitiligo)
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).

  o NOTE: Procedures such as a percutaneous biopsy, pleural catheter insertion, placement of a central venous catheter or other minor procedures are permitted.
* Uncontrolled or significant cardiovascular disease, including the following:
* Evidence of prolongation of QT/QTc interval (e.g., repeated episodes of QT corrected for heart rate using Fridericia's method [QTcF] >470 ms). Electrocardiogram must be registered at rest. For any ECG assessment, if the initial ECG shows a prolonged QTc, then two additional ECGs will be obtained, resulting in three specimens taken after a space of 1 minute, and the mean of the 3 ECGs will be used to determine eligibility and for grading of TRAEs.
* Myocardial infarction within 6 months prior to screening o Uncontrolled angina pectoris within 6 months prior to screening o New York Heart Association (NYHA) Class 3 or 4 congestive heart failure
* Uncontrolled hypertension (resting systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)
* Have a known hypersensitivity to any of the components of or known hypersensitivity to either the study drug itself or any of the inactive ingredients in the study drug product.
* Known liver cirrhosis.
* Uncontrolled active infection requiring IV antibiotic, antiviral, or anti-fungal medications within 14 days prior to initiation of study treatment.

  o Infections controlled on concurrent anti-microbial agents and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Congenital or acquired immunodeficiency, including patients with known history or infection with human immunodeficiency virus (HIV).

  o NOTE: HIV-positive patients who are taking anti-retroviral therapy are still ineligible due to potential PK interactions with valemetostat.
* Active tuberculosis
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test followed by a positive HBV RNA test within 28 days prior to the first dose of study drug. Hepatitis B testing (HBV surface antigen and core antibody) is required only if not done previously.

  o Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening, are eligible for the study.
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test within 28 days prior to the first dose of study drug. Hepatitis C testing (HCV antibody) is required only if not done previously.

  o The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Prior malignancy, active within the previous 3 years, except for locally curable cancer that is currently considered as cured or successfully resected, such as basal or squamous cell carcinoma, superficial bladder cancer, gastric cancer or carcinoma in situ of the prostate, cervix, or breast.
* Female patients who have a positive serum pregnancy test during screening or a positive urine pregnancy test on Day 1 before first dose of study drug.
* Female patients who are lactating and/or plan to breastfeed during the study treatment or at any point leading up to and including 6 months after the last study drug dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determine Phase II dose (RP2D) | 1 year
  The Common Terminology Criteria for Adverse Events (CTCAE) 5.0 will be used to determine all adverse events and dose-limiting toxicities.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  The Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria will be used to determine progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm